CLINICAL TRIAL: NCT06077474
Title: Validation and Reliability of the Turkish Version of the UCLA Posttraumatic Stress Disorder (PTSD) Reaction Index (RI) for The Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 Self Report for Children and Adolescents
Brief Title: Validation of the Turkish Version of PTSD-RI-5
Status: Completed | Type: Observational
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Melek Ince, MD, Dr. Behcet Uz Children's Hospital
Other Study IDs: 38583858
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Post-Traumatic Stress Disorder in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PTSD QUESTIONNAIRES: The group is anticipated to consist of in 155 patients who have been exposed to traumatic events.
  Interventions: Other: Testing the the DSM-5 UCLA Posttraumatic Stress Disorder Reaction Index Self-Report Scale for Children and Adolescents (PTSD-RI-5)

INTERVENTIONS:
Other: Testing the the DSM-5 UCLA Posttraumatic Stress Disorder Reaction Index Self-Report Scale for Children and Adolescents (PTSD-RI-5) — Administer the DSM-5 PTSD-RI-5 scale in 155 patients with exposed to traumatic events.
  Other Names: Severity of Post-Traumatic Stress Symptoms -Child aged 11-17 Post-Traumatic Stress Disorder National Stressful Events Survey Short Form (NSESSS)

SUMMARY:
The aim of this study is to investigate the adaptation and validity of the DSM-5 PTSD-RI -5 scale in patients who have been exposed to traumatic events. Thus, a scale useful for the diagnosis and follow-up of PTSD will be presented to the Turkish population.

DETAILED DESCRIPTION:
Children worldwide are at risk of experiencing psychological trauma. In addition, one in every four children experiences major traumatic events such as domestic, school, or social violence, abuse, vehicle accidents, serious medical diseases, terrorist incidents, and war. These difficult experiences increase the incidence of post-traumatic stress disorder in children. It is reported that approximately 30% of children who have been exposed to trauma develop post-traumatic stress disorder. Although it is sometimes difficult to diagnose post-traumatic stress disorder, it is important to detect symptoms of PTSD in children and adolescents early. Many internalizing and externalizing symptoms occur in PTSD; There may be separation anxiety, shame, guilt, low tolerance, overstimulation, impulsivity, outbursts of anger, hostility, defiance, aggression, irritability, and mood changes. Therefore, early evaluation of trauma experience and post-traumatic symptoms in children and adolescents seems important.

ELIGIBILITY:
Inclusion Criteria:

* Being a child or adolescent between the ages of 11-17
* To have experience a traumatic event in the past
* To have cognitive capacity to understand and complete the survey.

Exclusion Criteria:

-

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and Adolescents aged 11 and 17 with exposed to traumatic events
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Reliability of PTSD-RI-5 | Baseline
  Internal consistency will be tested with Cronbach Alpha coefficient. Test-retest reliability will be tested with intraclass correlation coefficient (ICC).
Reliability of PTSD-RI-5 | At the end of the 2nd week of study
  Test-retest reliability will be tested with intraclass correlation coefficient (ICC).
Correlation between the PTSD-RI-5 and Post-Traumatic Stress Disorder National Stressful Events Survey Short Form | Baseline
  The Spearman Correlation Analysis will be used for the correlation between between the PTSD-RI-5 and Post-Traumatic Stress Disorder National Stressful Events Survey Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Fatma S Durak, MD, Study Chair — Dr. Behcet Uz Children's Hospital
Locations (1):
- Dr. Behcet Uz Pediatric Diseases And Surgery Training And Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Campo-Arias A, Oviedo HC. [Psychometric properties of a scale: internal consistency]. Rev Salud Publica (Bogota). 2008 Nov-Dec;10(5):831-9. doi: 10.1590/s0124-00642008000500015. Spanish. PMID 19360231
- [Result] Costello EJ, Erkanli A, Fairbank JA, Angold A. The prevalence of potentially traumatic events in childhood and adolescence. J Trauma Stress. 2002 Apr;15(2):99-112. doi: 10.1023/A:1014851823163. PMID 12013070
- [Result] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Result] Dykman RA, McPherson B, Ackerman PT, Newton JE, Mooney DM, Wherry J, Chaffin M. Internalizing and externalizing characteristics of sexually and/or physically abused children. Integr Physiol Behav Sci. 1997 Jan-Mar;32(1):62-74. doi: 10.1007/BF02688614. PMID 9105915
- [Result] Yalin Sapmaz S, Ergin D, Ozek Erkuran H, Sen Celasin N, Ozturk M, Karaarslan D, Koroglu E, Aydemir O. Validity and Reliability of the Turkish Version of the DSM-5 Posttraumatic Stress Symptom Severity Scale-Child Form. Noro Psikiyatr Ars. 2017 Sep;54(3):205-208. doi: 10.5152/npa.2017.15913. Epub 2016 Sep 1. PMID 29033631
- [Result] Laor N, Wolmer L, Kora M, Yucel D, Spirman S, Yazgan Y. Posttraumatic, dissociative and grief symptoms in Turkish children exposed to the 1999 earthquakes. J Nerv Ment Dis. 2002 Dec;190(12):824-32. doi: 10.1097/00005053-200212000-00004. PMID 12486370
- [Result] Tsang S, Royse CF, Terkawi AS. Guidelines for developing, translating, and validating a questionnaire in perioperative and pain medicine. Saudi J Anaesth. 2017 May;11(Suppl 1):S80-S89. doi: 10.4103/sja.SJA_203_17. PMID 28616007
- [Result] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Result] Kaplow JB, Rolon-Arroyo B, Layne CM, Rooney E, Oosterhoff B, Hill R, Steinberg AM, Lotterman J, Gallagher KAS, Pynoos RS. Validation of the UCLA PTSD Reaction Index for DSM-5: A Developmentally Informed Assessment Tool for Youth. J Am Acad Child Adolesc Psychiatry. 2020 Jan;59(1):186-194. doi: 10.1016/j.jaac.2018.10.019. Epub 2019 Apr 3. PMID 30953734
- [Result] Tavakol M, Dennick R. Making sense of Cronbach's alpha. Int J Med Educ. 2011 Jun 27;2:53-55. doi: 10.5116/ijme.4dfb.8dfd. No abstract available. PMID 28029643
- [Result] Schober P, Boer C, Schwarte LA. Correlation Coefficients: Appropriate Use and Interpretation. Anesth Analg. 2018 May;126(5):1763-1768. doi: 10.1213/ANE.0000000000002864. PMID 29481436